CLINICAL TRIAL: NCT03114306
Title: Implementation of a Fast-track Knee Arthroplasty Concept: a Randomized, Controlled, Open Clinical Trial
Brief Title: Evaluation of a Fast-track Knee Arthroplasty Concept
Acronym: KneeOptOut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Sascha Treskatsch, Head of department, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KneeOptOut
Record Dates: First submitted 2017-03-27; First posted 2017-04-14 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Knee Arthropathy; Postoperative Pain; Postoperative Complications
Keywords: ERAS; pain; knee arthroplasty; joint pain; regional anaesthesia
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications; Pain; Arthralgia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and treating physicians are different in this trial, that means, the assessor of primary study endpoint will be blinded regarding group allocation. Patients receive either regional-anaesthesiological catheters preoperatively or are treatet with local infiltration technique perioperatively. For the purpose of this trial is would not be feasable to perform sham regional-anaesthesiological procedures and blinding of the treating physisican will not be possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- local infiltration analgesia (Experimental): Patient receive an infiltration of local anaesthetics around the knee to achieve maximal distal block of nerve fibres. Infiltration is performed directly after knee replacement and during weaning of general anaesthesia.
  Interventions: Procedure: local infiltration analgesia
- Regional anaesthesia (Active Comparator): Patients receive a combined anaesthesia with a regional-anaesthesiological catheter placed close to the distal Nervus saphenus and a single shot anaesthesia of Nervus ischiadicus using local anaesthetics (regional-anaesthesiological catheter analgesia).
  Interventions: Procedure: regional-anaesthesiological catheter analgesia

INTERVENTIONS:
Procedure: local infiltration analgesia — Patient receive an infiltration of local anaesthetics around the knee directly after total knee replacement for postoperative pain control.
  Other Names: LIA technique
  Arms: local infiltration analgesia
Procedure: regional-anaesthesiological catheter analgesia — Patients receive a single shot nerve block of the proximal Nervus ischiadicus and a catheter placed closed to the Nervus saphenus for perioperative pain control using ultrasound guided techniques.
  Arms: Regional anaesthesia

SUMMARY:
Mobilisation following knee arthroplasty is an important aspect to achieve early and enhanced recovery after surgery and sufficient joint function. Analgesia is a crucial therapeutic element in this context. This RCT evaluates two analgetic regimens for patients undergoing primary total knee-replacement to assess impact on postoperative recovery.

DETAILED DESCRIPTION:
Mobilisation following knee arthroplasty is important for patients to achieve early and enhanced recovery after surgery and sufficient joint function. Analgesia is a crucial therapeutic element in this context. There is evidence that regional- anaesthesiological catheter techniques are very efficient to control pain postoperatively. On the other hand, motoric function may be reduced due to nerve blocks depending on location and concentration of drug used. Local infiltration of the knee during surgery is an alternative component in pain management that may reduce impaired motor function and allow early mobilisation of patients. However, currently it is not known which analgesia technique provides optimal pain control paralleled with sufficient motor function. Against this background, this RCT evaluates two analgesia regimens for patients undergoing primary total knee-replacement to assess impact on postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective, primary knee joint replacement in combined general anaesthesia

Exclusion Criteria:

* heart insufficiency NYHA >2
* liver insufficiency > CHILD B
* evidence of diabetic polyneuropathy
* severe adipositas BMI >40
* patients < 18 years
* pregnancy
* in case of police custody
* participation in a paralleled interventional RCT in a time frame of 30 days
* chronic opioid therapy >3 months before scheduled surgery
* allergy against medication required for surgery or anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
time to first mobilisation (standing) | up to 48h postoperatively
  time from end of surgery until patients is able to stand

SECONDARY OUTCOMES:
patients satisfaction (11-point likert scale) | up to 7 days postoperatively
  global satisfaction of patients
time to first mobilisation (walking) | up to 7 days postoperatively
  time from end of surgery until patients is able to walk
complications | up to 7 days postoperatively
  complications during perioperative care process (e.g. thrombosis, re-operation, infection)
time to achieve full joint mobility | up to 7 days postoperatively
  time to achieve full joint mobility (0/0/90°)
pain intensity of patients (11-point likert visual analogue scale) measured 3 times daily (mean) | up to 7 days postoperatively
  mean pain intensity of patients
rescue pain medication | up to 7 days postoperatively
  number of patients requiring rescue pain medication
pain medication perioperatively | up to 7 days postoperatively
  pain medication perioperatively (e.g. NSAIDs, opioids, con-analgetics)
time to discharge | up to 14 days postoperatively
  time to discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Treskatsch, Prof., Principal Investigator — Charite University Berlin, Department of anaesthesia
Locations (1):
- Charité University Berlin (CCM), Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Individual requests to analyse data are to be evaluated by local data safety authorities

REFERENCES:
- [Background] Rostlund T, Kehlet H. High-dose local infiltration analgesia after hip and knee replacement--what is it, why does it work, and what are the future challenges? Acta Orthop. 2007 Apr;78(2):159-61. doi: 10.1080/17453670710013627. No abstract available. PMID 17464601
- [Background] Peters CL, Shirley B, Erickson J. The effect of a new multimodal perioperative anesthetic regimen on postoperative pain, side effects, rehabilitation, and length of hospital stay after total joint arthroplasty. J Arthroplasty. 2006 Sep;21(6 Suppl 2):132-8. doi: 10.1016/j.arth.2006.04.017. PMID 16950075
- [Result] Kastelik J, Fuchs M, Kramer M, Trauzeddel RF, Ertmer M, von Roth P, Perka C, Kirschbaum SM, Tafelski S, Treskatsch S. Local infiltration anaesthesia versus sciatic nerve and adductor canal block for fast-track knee arthroplasty: A randomised controlled clinical trial. Eur J Anaesthesiol. 2019 Apr;36(4):255-263. doi: 10.1097/EJA.0000000000000929. PMID 30562225
- [Result] Borck M, Wandrey JD, Hoft M, Kastelik J, Perka C, Tafelski S, Treskatsch S. Local infiltration analgesia versus peripheral nerve block anaesthesia in total knee arthroplasty: a pharmaco-economic comparison. BMC Anesthesiol. 2022 Mar 25;22(1):80. doi: 10.1186/s12871-022-01620-w. PMID 35337268